CLINICAL TRIAL: NCT00564798
Title: Shapedown BC Program Evaluation
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H07-00243
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Obesity
Keywords: protocoladolescents; children; health behaviours/attitudes; weight loss/management; program evaluation
MeSH Terms: conditions — Obesity; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Study Group
- 2: Control Group

SUMMARY:
Shapedown BC is being implemented at a single centre (BC's Children's Hospital). We will use the data routinely collected by the Shapedown program and evaluate the effect of the program and whether any changes are sustained for up to 2 years. A group of subjects who expressed interest in the program but ultimately decided not to participate will be used as a reference group.

DETAILED DESCRIPTION:
With the increase in obesity among children and adolescents in Canada, there is a commensurate rise in the incidence of type 2 diabetes (T2D), and the age at which it is appearing is getting lower. Reversing obesity is a critical primary intervention for the prevention of the development of T2D in children/adolescents. Achieving long-term weight change has proven to be very difficult, particularly for children. The Shapedown program is a well-structured but resource-intensive program for weight management in children and adolescents. Like many obesity intervention programs, its efficacy has not been evaluated. If it is shown to have long term impact on obesity, and thus reduce the incidence of T2D and the demand on the health care system for other co-morbidities of obesity, the costs are likely warranted. However, if Shapedown is not efficacious at reversing obesity or the physiologic markers for its complications, the high demand on health care resources may not be warranted.

Hypothesis The Shapedown treatment group will have a reduction in Body Mass Index (BMI) of 0.75 kg/m2 at 3 months compared to baseline evaluation and this reduction will be sustained for 12 and 24 months.

Primary Objective To determine whether Shapedown BC is efficacious at reducing BMI by 0.75 kg/m2 at the completion of the 10 week treatment program (3 month assessment)

Secondary Objectives:

1. To determine whether the reduction in BMI achieved at 3 months can be sustained at 6, 12, 18 and 24 months after the Shapedown intervention.
2. To describe changes in BMI in a Natural History group (those choosing not to participate in Shapedown) at 3, 6, 12, 18, 24 months.
3. To perform a process evaluation of the Shapedown program with respect to participation, satisfaction and attrition.
4. To perform an exploratory analysis of the psychological assessments of the Shapedown treatment group at the end of the program, 3 and 12 months post-intervention compared to baseline.
5. To evaluate changes in physical fitness in the Shapedown treatment group at the end of Shapedown program, 3 and 12 months post intervention compared to baseline.

Research Design The program will be evaluated by following a prospective cohort of those treated through the Shapedown program, with the additional component of a "Natural History",non-participant group.

Relevance Obesity is the primary risk factor for the development of T2D.

Outcome/Impact This study provides critical data on the efficacy of Shapedown as a weight management program as well as its effect on changing insulin resistance in children. We will also gain important epidemiological information on the co-morbidities present in obese children. We will also gain knowledge on the reasons certain families decline to participate, barriers to treatment, as well as the natural history of weight gain in the non-participant group.

ELIGIBILITY:
Inclusion Criteria:

All children/families meeting the criteria for the the Shapedown BC program (families and children referred to the Shapedown program).

1. Age 6-18 years inclusive
2. Body mass index greater than or equal to the 95th percentile standardized for age and sex or Body mass index greater than or equal to 85th percentile but less than 95th percentile with co-morbidities such as hypertension, IGT, or type 2 diabetes, PCOS, dyslipidemia, and NASH.
3. Parents or primary care givers/guardians willing to attend the two intake sessions with the expectation that they will be required to participate in the entire program.

Exclusion Criteria:

Any child NOT referred to the Shapedown program.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A prospective evaluation study of the "Shapedown" BC program (Canada) for children aged 6-18 years.
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Panagiotopoulos, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada